CLINICAL TRIAL: NCT06892470
Title: Assessment of Postoperative Visual Outcomes in Highly Myopic Patients Implanted with Different Intraocular Lenses
Brief Title: Visual Quality of Cataract Patients with High Myopia After Implantation of Different Intraocular Lenses
Status: Active, not recruiting | Type: Observational
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Yune Zhao, Vice president of Eye Hospital of Wenzhou Medical University, Wenzhou Medical University
Other Study IDs: H2025-015-K-14-04
Record Dates: First submitted 2025-03-21; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- TNF Group:: Implantation of PanOptix trifocal IOL
  Interventions: Other: No intervention
- ZFR Group:: Implantation of Tecnis Symfony ZFR00 extended depth of focus IOL (Johnson & Johnson)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This prospective study aims to compare the visual outcomes following the implantation of two different types of multifocal intraocular lenses (IOLs) in highly myopic patients. The study will evaluate visual quality, refractive outcomes, and patient satisfaction using various visual assessment techniques and subjective satisfaction surveys.

ELIGIBILITY:
Inclusion Criteria:

* 1: Patients are older than 18 years

  2: The axial length (AL) measured by IOLMaster 700 is ≥26 mm

  3: No anterior or posterior segment pathology that could potentially compromise visual potential (such as glaucoma, myopic traction maculopathy, corneal leukoma, etc.).

  4: Able to understand, cooperate, and complete all follow - ups

Exclusion Criteria:

* 1: History of amblyopia

  2: Retinal detachment in the same eye or the fellow eye

  3: Presence of multiple peripheral retinal degenerative changes

  4: History of previous ocular surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals who undergo micro-incision cataract surgery and implantation of targeted intraocular lenses at the Hangzhou Branch of Wenzhou Medical University Eye Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Defocus Curve | Three months after operation
  The defocus curve is a tool used to assess visual acuity, particularly widely applied in evaluating the performance of presbyopia-correcting intraocular lenses (IOLs). Its principle involves placing a series of positive and negative lenses of varying diopters in front of the patient's eyes to simulate different distances from near to far, thereby assessing the patient's visual acuity (VA) at each simulated distance.
Visual Questionnaire | Three months after operation
  A visual questionnaire is a tool used to assess patients' visual function and quality of life. It typically includes a series of questions covering various aspects such as visual acuity at different distances (e.g., distance, intermediate, and near vision), dependency on glasses, and the impact of vision on the quality of life. By using a visual questionnaire, one can understand the actual visual experience and satisfaction of patients after the implantation of an intraocular lens.

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmology and Optometry Hos, Hanzhou, Zhejian, China

IPD SHARING:
Plan to Share IPD: No